CLINICAL TRIAL: NCT02625363
Title: Water Intake and Glycemic Response : Preliminary Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nutrifood Research Center, Jakarta, Indonesia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Nutrifood
Record Dates: First submitted 2015-11-16; First posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: Glycemic Index; Water Intake; Glycemic Response
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Glucose Ref - Std (Experimental): 250 ml glucose solution with 50 gram available carbohydrate per serving, used as reference
  Interventions: Other: Glucose Ref - Std
- Glucose Ref and 450 ml water (Experimental): 250 ml glucose solution with 50 gram available carbohydrate per serving. Sample was consumed with additional water intake @150 ml at 45, 75, and 105 minutes after meal consumption
  Interventions: Other: Glucose Ref and 450 ml water
- White Bread with 250 ml water (Experimental): White bread with 50 gram available carbohydrate was consumed with 250 ml water immediately after meal consumption
  Interventions: Other: White Bread with 250 ml water
- White Bread and 700 ml water (Experimental): White bread with 50 gram available carbohydrate was consumed with 250 ml water immediately after meal consumption. Moreover, subjects given additional water intake @150 ml at 45, 75, and 105 minutes after meal consumption
  Interventions: Other: White Bread and 700 ml water
- White Bread with 125 ml water (twice) (Experimental): Sample consumed with 125 ml water immediately after meal consumption, and additional 125 ml water after 60 minutes
  Interventions: Other: White Bread with 125 ml water (twice)

INTERVENTIONS:
Other: Glucose Ref - Std — First, fasting blood glucose was measured. Then, subjects consumed the glucose sample in 5-10 minutes and blood sugar level were measured at 0', 15', 30', 45', 60', 90', and 120'
  Arms: Glucose Ref - Std
Other: Glucose Ref and 450 ml water — First, fasting blood glucose was measured. Then, subjects consumed the glucose sample in 5-10 minutes. Subjects given additional 150 ml water at 45, 75, and 105 minutes and blood sugar level were measured at 0', 15', 30', 45', 60', 90', and 120
  Arms: Glucose Ref and 450 ml water
Other: White Bread with 250 ml water — First, fasting blood glucose was measured. Then, subjects consumed the samples in 10-15 minutes and blood sugar level were measured at 0', 15', 30', 45', 60', 90', and 120'
  Arms: White Bread with 250 ml water
Other: White Bread and 700 ml water — Sample consumed with 250 ml water immediately after meal consumption, and additional 150 ml water at 45, 75, and 105 minutes.
  First, fasting blood glucose was measured. Then, subjects consumed the samples in 10-15 minutes and blood sugar level were measured at 0', 15', 30', 45', 60', 90', and 120'
  Arms: White Bread and 700 ml water
Other: White Bread with 125 ml water (twice) — Sample consumed with 125 ml water immediately after meal consumption, and additional 125 ml water after 60 minutes
  First, fasting blood glucose was measured. Then, subjects consumed the samples in 10-15 minutes and blood sugar level were measured at 0', 15', 30', 45', 60', 90', and 120'
  Arms: White Bread with 125 ml water (twice)

SUMMARY:
Glycemic index concept is widely used to determine impact of a food to blood glucose. Several studies showed that water content and intake after meal may influence glycemic response of the meal and thus have an effect on the result of GI measurement. Currently these studies found conflicting results. Therefore, this study aims to determine whether water intake, specifically after meal, may influence the glycemic response and glycemic index value of the meal.

DETAILED DESCRIPTION:
Glycemic index methods are performed according to Food and Agricultural Organization/WHO recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-40 years
* fasting blood glucose 70-99 mg/dL
* Indonesians

Exclusion Criteria:

* having diabetes
* smoking
* if women, pregnant or lactating
* being allergic to food used in this study
* having gastrointestinal disturbance
* in regular medication
* refusal to sign the consent form

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
2 h postprandial blood glucose level (Glycemic Response) | fasting 0 min, 15 min, 30 min, 45 min, 60 min, 90 min, 120 min
Glycemic index value of meal (white bread) | fasting 0 min, 15 min, 30 min, 45 min, 60 min, 90 min, 120 min
  The glycemic index is a calculated from measurements of area under the glucose curve after the food is eaten, divided by the corresponding area after the control food is eaten. The value is multiplied by 100 to represent a percentage of the reference food.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Yolanda, SSi, Principal Investigator — Nutrifood Research Center; Astri Kurniati, MAppSc, Study Chair — Nutrifood Research Center; Lina Antono, MSc, Principal Investigator — Nutrifood Research Center
Locations (1):
- PT Nutrifood Indonesia, Jakarta, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Carbohydrates in human nutrition. Report of a Joint FAO/WHO Expert Consultation. FAO Food Nutr Pap. 1998;66:1-140. No abstract available. PMID 9743703
- [Background] Young KWH, Wolever TMS. Effect of volume and type of beverage consumed with a standard test meal on postprandial blood glucose responses. Nutrition Research 18(11): 1857-1863, 1998
- [Background] Torsdottir I, Andersson H. Effect on the postprandial glycaemic level of the addition of water to a meal ingested by healthy subjects and type 2 (non-insulin-dependent) diabetic patients. Diabetologia. 1989 Apr;32(4):231-5. doi: 10.1007/BF00285289. PMID 2759361
- [Background] Gregersen S, Rasmussen O, Winther E, Hermansen K. Water volume and consumption time: influence on the glycemic and insulinemic responses in non-insulin-dependent diabetic subjects. Am J Clin Nutr. 1990 Sep;52(3):515-8. doi: 10.1093/ajcn/52.3.515. PMID 2203255